CLINICAL TRIAL: NCT00785980
Title: A One-Directional, Open-Label Drug Interaction Study to Investigate the Effects of Multiple-Dose Ciprofloxacin HCl on the Single-Dose Pharmacokinetics of Quinine in Healthy Volunteers
Brief Title: Drug - Drug Interaction Study of Quinine Sulfate and Ciprofloxacin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-001-08-1027
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Results first posted 2009-10-21 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: quinine sulfate; ciprofloxacin; drug interactions; cytochrome p450; male; female; adult; pharmacokinetics
MeSH Terms: interventions — Quinine; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quinine Sulfate (Active Comparator): Baseline quinine sulfate pharmacokinetics
  Interventions: Drug: Quinine Sulfate Capsules 324 mg
- Quinine Sulfate with Ciprofloxacin (Experimental): Quinine sulfate pharmacokinetics in the presence of steady state ciprofloxacin
  Interventions: Drug: Ciprofloxacin 500 mg; Drug: Quinine Sulfate Capsules 324 mg

INTERVENTIONS:
Drug: Quinine Sulfate Capsules 324 mg — A single dose of quinine sulfate (2 x 324 mg capsules) administered on the morning of Day 1 after an overnight fast of at least 10 hours.
  Other Names: Qualaquin®
  Arms: Quinine Sulfate
Drug: Ciprofloxacin 500 mg — A single dose of quinine sulfate (2 x 324 mg capsules) co-administered with a single dose of ciprofloxacin (1 x 500 mg tablet) in the morning on Day 11 after an overnight fast of at least 10 hours.
  Other Names: Cipro®
  Arms: Quinine Sulfate with Ciprofloxacin
Drug: Quinine Sulfate Capsules 324 mg — A single dose of quinine sulfate (2 x 324 mg capsules) co-administered with a single dose of ciprofloxacin (1 x 500 mg tablet) in the morning on Day 11 after an overnight fast of at least 10 hours.
  Other Names: Qualaquin®
  Arms: Quinine Sulfate with Ciprofloxacin

SUMMARY:
Ciprofloxacin is moderate inhibitor of cytochrome P450 1A2 (CYP1A2), one of the enzymes responsible for the metabolism of quinine. This study will evaluate the effect of ciprofloxacin-related inhibition of CYP1A2 on the pharmacokinetics of quinine sulfate.

DETAILED DESCRIPTION:
Ciprofloxacin is moderate inhibitor of cytochrome P450 1A2 (CYP1A2), one of the enzymes responsible for the metabolism of quinine. This study will evaluate the effect of ciprofloxacin-related inhibition of CYP1A2 on the pharmacokinetics of quinine sulfate. In the morning on study Day 1 after a fast of at least 10 hours, twenty-four healthy, non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 will be given one oral dose of quinine sulfate (2 x 324 mg capsules). Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 36 hours post-dose at times sufficient to adequately define the pharmacokinetics of quinine sulfate. A 7-day washout period will be completed after the first dose of quinine sulfate on Day 1. Beginning at 07:45 am on Day 8 and continuing through Day 10, all subjects will return to the clinic for non-confined dosing of ciprofloxacin (1 x 500 mg tablet) every 12 hours. Administered ciprofloxacin doses on these days will not be in a fasted state. At 07:45 am on Day 11 after a fast of at least 10 hours, all study participants will receive a co-administered single oral dose of quinine sulfate (2 x 324 mg capsules) and ciprofloxacin (1 x 500 mg tablet). A final dose of ciprofloxacin (1 x 500 mg tablet) will be administered 12 hours later. Blood samples will be drawn from all participants before dosing and for 36 hours post-dose at times sufficient to adequately define the pharmacokinetics of quinine sulfate. Fasting will continue for 4 hours following the co-administered dose of quinine sulfate and ciprofloxacin. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Seated blood pressure and pulse will be measured pre-dose and at 1, 2 and 3 hours post-dose on Days 1 and 11. An electrocardiogram (ECG) will be done pre-dose and at 1, 2 and 4 hours post-dose on Days 1 and 11. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age
* Non-smoking
* Non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures)
* Body mass index (BMI)between 18 and 32
* Medically healthy on the basis of medical history and physical examination
* Hemoglobin > or = to 11.5 g/dL
* Completion of the screening process within 28 days prior to dosing
* Provision of voluntary written informed consent

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study
* Drug allergies to mefloquine or quinidine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, PharmD, Principal Investigator — PRACS Institute, Ltd.

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four (24) healthy, non-smoking, adult male and female volunteers from the community at large were enrolled.
Pre-assignment Details: Thirty-nine (39) subjects were screened. Four (4) did not meet eligibility criteria, nine (9) had a schedule conflict prior to Period I check-in, and two (2) transferred to another study.
Groups:
- Quinine Alone, Ciprofloxacin Alone, Quinine With Ciprofloxacin: All subjects received a single dose of quinine sulfate (2 x 324 mg capsules) on Day 1 following an overnight fast of at least 10 hours. After a 7-day washout period, beginning on the morning of Day 8 subjects received a dose of ciprofloxacin (1 x 500 mg tablet) twice a day for 4 days. On Day 11 in the morning, subjects received a single dose of quinine sulfate (2 x 324 mg capsules) co-administered with a single dose of ciprofloxacin (1 x 500 mg tablet). On Day 11 in the evening, the final dose of ciprofloxacin (1 x 500 mg tablet) was administered.
Period: Quinine Sulfate Alone
Arm/Group | Quinine Alone, Ciprofloxacin Alone, Quinine With Ciprofloxacin
Started | 24
Completed | 24
Not Completed | 0
Period: 7 Day Washout Period
Arm/Group | Quinine Alone, Ciprofloxacin Alone, Quinine With Ciprofloxacin
Started | 24
Completed | 21
Not Completed | 3
Not completed — Protocol Violation | 3
Period: Ciprofloxacin Alone
Arm/Group | Quinine Alone, Ciprofloxacin Alone, Quinine With Ciprofloxacin
Started | 21
Completed | 21
Not Completed | 0
Period: Quinine Sulfate With Ciprofloxacin
Arm/Group | Quinine Alone, Ciprofloxacin Alone, Quinine With Ciprofloxacin
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Quinine Alone, Ciprofloxacin Alone, Quinine With Ciprofloxacin
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.9 (7.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration(Cmax)
Description: The maximum or peak concentration that the drug reaches in the plasma.
Time Frame: Serial pharmacokinetic blood samples for quinine sulfate collected on Days 1 and 11 before dosing and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 36 hours post-dose.
Population: Pharmacokinetic analyses are based on twenty-one (21) subjects who successfully completed the study. Three (#3) subjects were dropped by the sponsor due to protocol violation.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Quinine Sulfate Alone: On Day 1 in the morning, after a fast of at least 10 hours, all subjects received a single dose of quinine sulfate (2 x 324 mg capsules) followed by a 7-day washout period.
- Quinine Sulfate With Ciprofloxacin: On Day 11 in the morning, after a fast of at least 10 hours, all subjects received a single dose of quinine sulfate (2 x 324 mg capsules) co-administered with a single dose of ciprofloxacin (1 x 500 mg).
Arm/Group | Quinine Sulfate Alone | Quinine Sulfate With Ciprofloxacin
Number analyzed (Participants) | 21 | 21
ng/mL | 4,240.65 (1,162.25) | 4,521.20 (1,122.28)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve beginning from the first dose (time 0) to the last measurable concentration (time t), as calculated by the linear trapezoidal method.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Quinine Sulfate Alone | Quinine Sulfate With Ciprofloxacin
Number analyzed (Participants) | 21 | 21
ng-hr/mL | 63,415.67 (16,009.17) | 68,572.17 (18,922.82)

3. Primary Outcome: Area Under the Concentration Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)].
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞)was calculated as the sum of the AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Population: Pharmacokinetic analyses are based on 20 subjects out of the 21 subjects who completed the study. One value was determined to be unreliable and was not used.
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Quinine Sulfate Alone | Quinine Sulfate With Ciprofloxacin
Number analyzed (Participants) | 20 | 20
ng-hr/mL | 67,694.99 (15,644.74) | 77,439.24 (26,083.49)

ADVERSE EVENTS:
Description: 24 subjects were enrolled in this study. Several subjects dropped out of the study prior to receiving all interventions. 24 subjects were administered Quinine sulfate, 21 subjects were administered Ciprofloxacin and 18 subjects were co-administered Quinine Sulfate and Ciprofloxacin.
Groups:
- Quinine Sulfate Alone: On Day 1 in the morning, after a fast of at least 10 hours, all subjects received a single dose of quinine sulfate (2 x 324 mg capsules) followed by a 7-day washout period. On Day 11 in the morning, all subjects received a single dose of quinine sulfate (2 x 324 mg capsules) co-administered with a single dose of ciprofloxacin (1 x 500 mg tablet) following an overnight fast of 10 hours.
- Ciprofloxacin Alone: Beginning on Day 8 in the morning and continuing through Day 11 in the evening, all subjects received a dose of ciprofloxacin (1 x 500 mg tablet) twice daily for a total of 8 doses.
- Quinine Sulfate With Ciprofloxacin: On Day 11 in the morning, all subjects received a dose of quinine sulfate (2 x 324 mg capsules) co-administered with a dose of ciprofloxacin (1 x 500 mg tablet) after an overnight fast of at least 10 hours.
Arm/Group | Quinine Sulfate Alone | Ciprofloxacin Alone | Quinine Sulfate With Ciprofloxacin
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21 | 0/18
Other Adverse Events (participants affected / at risk) | 9/24 | 1/21 | 3/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quinine Sulfate Alone (N=24) | Ciprofloxacin Alone (N=21) | Quinine Sulfate With Ciprofloxacin (N=18)
Ear discomfort (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days